CLINICAL TRIAL: NCT05676294
Title: The Impact of Pre-operative Olanzapine on Quality of Recovery-40 Scores After Discharge From Ambulatory Surgery
Brief Title: The Impact of Preoperative Olanzapine on Quality of Recovery After Discharge From Ambulatory Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Jaime B. Hyman, MD, Associate Professor of Anesthesiology, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2000033786; No NIH funding (Other: 12.06.23)
Record Dates: First submitted 2022-12-21; First posted 2023-01-09 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: olanzapine; placebo-controlled; nausea; vomiting; ambulatory surgery procedures; antiemetic; general anesthesia
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olanzapine (Experimental): olanzapine oral tablet, 5mg, once prior to surgery
  Interventions: Drug: Olanzapine
- Placebo (Placebo Comparator): placebo oral tablet once prior to surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olanzapine — 5 mg of oral olanzapine one hour prior to ambulatory surgery
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Placebo — oral matched placebo one hour prior to ambulatory surgery
  Arms: Placebo

SUMMARY:
The primary objective of this phase 2 randomized controlled trial is to determine whether the pre-operative administration of olanzapine (5 mg PO) improves quality of recovery (assessed by the Quality of Recovery-40 (QoR-40) survey) on postoperative day 1 in patients having ambulatory surgery with general anesthesia.

The secondary objectives of this study are to determine whether there are differences in quality of recovery on postoperative day 2, presence of post-discharge nausea, presence of severe post-discharge nausea, recovery room length of stay and opioid consumption in patients who receive the study drug versus placebo.

DETAILED DESCRIPTION:
Up to 37% of patients undergoing ambulatory surgery experience postdischarge nausea and vomiting (PDNV), and PDNV represents a major barrier to improving a patient's quality of recovery. Because olanzapine has been shown to be an effective drug for PDNV prevention, but carries the risk of sedation, this study seeks to identify if the administration of olanzapine is an intervention that improves a patient's overall quality of recovery.

The study population includes women between 18 and 50 years-old who are undergoing ambulatory (outpatient) surgery at Yale New Haven Hospital. This represents the population that is most susceptible to post-discharge nausea and vomiting (PDNV) and is therefore most likely to benefit from an intervention that reduces PDNV to impact overall quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Female aged 18-50
* Scheduled to undergo ambulatory surgery under general anesthesia
* Access to smartphone device or computer with internet connection and has an email address

Exclusion Criteria:

* Non-English speaking
* Unable to swallow pills
* Current use of anti-psychotic medications
* History of allergy to olanzapine
* Pregnancy/Lactation
* Current use of antihypertensive medication
* Diabetes Mellitus
* Clinically significant cardiovascular disease defined as follows:

  1. Myocardial infarction or unstable angina within 6 months prior to the day of planned surgery.
  2. History of serious ventricular arrhythmia (i.e.: ventricular tachycardia or ventricular fibrillation) or cardiac arrhythmias requiring anti-arrhythmic medications, except for atrial fibrillation that is well controlled on anti-arrhythmic medication.
  3. New York Heart Association Class II or higher congestive heart failure.
  4. Postural hypotension or vasovagal syncope within 6 months of planned surgery.
* Hypotension on day of surgery, defined as a systolic blood pressure < 90mmHg
* Seizure disorder
* Clinically active prolactinoma
* Hepatic disease
* Narrow angle glaucoma
* Parkinson's disease
* Lewy body dementia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 384 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2025-12-06 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery-40 (QoR-40) survey to assess efficacy | post-operative day 1
  Quality of Recovery-40 (QoR-40) survey is a 40-item questionnaire that provides a global score across five dimensions: patient support, comfort, emotions, physical independence, and pain. The survey is scored on a 5-point Likert scale: for positive items: 1 = none of the time, 5 = all of the time; for negative items, the scoring was reversed. The QoR-40 has a possible score of 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).

SECONDARY OUTCOMES:
Quality of Recovery-40 (QoR-40) survey to assess efficacy | post-operative day 2
  Quality of Recovery-40 (QoR-40) survey is a 40-item questionnaire that provides a global score across five dimensions: patient support, comfort, emotions, physical independence, and pain. The survey is scored on a 5-point Likert scale: for positive items: 1 = none of the time, 5 = all of the time; for negative items, the scoring was reversed. The QoR-40 has a possible score of 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).
Nausea | post-operative day 1
  Presence of nausea on post-operative day 1 will be rated on a 0 to 10 numerical rating scale with 0 being "none" and 10 being "worst nausea imaginable"
Nausea | post-operative day 2
  Presence of nausea on post-operative day 2 will be rated on a 0 to 10 numerical rating scale with 0 being "none" and 10 being "worst nausea imaginable"
Severe post-discharge nausea | up to 24 hours post discharge
  Severe post-discharge nausea defined as any numerical rating > 3 on a 0-10 scale during the 24 hours after discharge
Recovery room length of stay | From surgery end time to recovery room discharge, up to 23 hours
  Recovery room length of stay in minutes
Recovery room opioid consumption | From surgery end time to recovery room discharge, up to 23 hours
  Recovery room opioid consumption in morphine milligram equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Hyman, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hyman JB, Park C, Lin HM, Cole B, Rosen L, Fenske SS, Barr Grzesh RL, Blank SV, Polsky SB, Hartnett M, Taub PJ, Palvia V, DeMaria S Jr, Ascher-Walsh C. Olanzapine for the Prevention of Postdischarge Nausea and Vomiting after Ambulatory Surgery: A Randomized Controlled Trial. Anesthesiology. 2020 Jun;132(6):1419-1428. doi: 10.1097/ALN.0000000000003286. PMID 32229754